CLINICAL TRIAL: NCT02300870
Title: Myocardial Perfusion Echocardiography to Detect Human Heart Transplant
Brief Title: Myocardial Perfusion Echocardiography to Detect Human Heart Transplant Rejection
Status: Terminated | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: General Electric (Industry)
Responsible Party: Principal Investigator, Michael Givertz, MD, Medical Director, Heart Transplant and Mechanical Circulatory Support, Brigham and Women's Hospital
Other Study IDs: BWHMG370000
Record Dates: First submitted 2014-11-17; First posted 2014-11-25 (Estimated); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Heart Transplantation
Keywords: Acute rejection, myocardial blood flow
MeSH Terms: interventions — FS 069

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Heart Transplant Rejection: Patients presenting with acute cellular rejection
  Interventions: Drug: Optison
- Heart Transplant Control: Patients presenting for routine office visit
  Interventions: Drug: Optison

INTERVENTIONS:
Drug: Optison — Echocardiogram with IV contrast
  Other Names: Echocontrast agent

SUMMARY:
The primary objective of this proposal is to show the efficacy of contrast enhanced ultrasonography in detecting heart transplant rejection in humans. The secondary objective is to demonstrate the efficacy of this technique in generating data which allow for the assessment of short and long term outcomes.

ELIGIBILITY:
Inclusion Criteria:

* All adult subjects (ages 18 to 75) who have undergone heart transplant at Brigham and Women's Hospital

Exclusion Criteria:

* hemodynamic instability (e.g., systolic blood pressure < 90 mmHg)
* atrial fibrillation with rapid ventricular response (e.g., heart rate > 120 bpm)
* premature atrial or ventricular complexes of a frequency that will not allow adequate echocardiographic assessment
* poor acoustic windows
* inability to provide informed consent
* any contraindication listed in the Optison package insert (i.e., history of an allergic reaction)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart Transplant patients
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2015-01; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Global and regional microvascular myocardial perfusion | Baseline
  Myocardial blood flow (dB/s)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Givertz, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No